CLINICAL TRIAL: NCT04066647
Title: Detection of miRNAs in HPA Axis Function in Healthy Subjects
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Interim analysis shows results opposite of hypothesized.
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Anat Ben-Shlomo, MD, Staff Physician, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro57715
Record Dates: First submitted 2019-07-24; First posted 2019-08-26 (Actual); Results first posted 2020-07-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Dexamethasone Effect on miRNA Profile in Healthy Humans
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dexamthesone (Experimental): Single arm study in which all healthy controls will receive 1 mg of dexamethasone intravenous (IV) injection.
  Interventions: Drug: Dexamethasone 4mg

INTERVENTIONS:
Drug: Dexamethasone 4mg — 1 mg IV dexamethasone will be pushed and miRNA levels will be checked at baseline just before injection and then at 15, 30, 45, and 60 minutes after injection.

SUMMARY:
The proposed study will test dexamethasone effect on miRNA profile in healthy humans. As our data indicate that miRNA levels change over time, the investigators will study the time course of miRNA response to 1 mg IV dexamethasone within 60 minutes after injection. Dexamethasone is used routinely in human subjects for the treatment of inflammatory conditions and as a diagnostic tool in the evaluation of excess cortisol secretion (Cushing's syndrome). For the latter, 1 mg dexamethasone is given orally at midnight. Oral formula absorption in the gut can range from 20 to 60 minutes due to the presence of food and other factors. IV administration will bypass this variability and ensure an accurate and reproducible time-course study. The investigators will compare miRNA expression before and after dexamethasone treatment. The investigators will follow miRNA expression dynamics over a 1-hour time course to identify peak expression levels and to correlate miRNA expression with circulating dexamethasone levels. Dexamethasone and miRNA levels will be checked at baseline just before injection and then at 15, 30, 45, and 60 minutes after injection. Dexamethasone level is taken to verify treatment and to correlate it with miRNA expression.

ELIGIBILITY:
Inclusion Criteria:

* Adults age ≥ 18

Exclusion Criteria:

* Pregnancy
* Presence of a disease that affects HPA axis function
* Current use of medications that affect cortisol secretion, such as opioid pain medication, anti-fungal agents, anti-epileptic agents, and glucocorticoids, including hydrocortisone, prednisone, dexamethasone, steroid-containing inhalers, and steroid injected into the joints
* History of adverse event related to use of glucocorticoids

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2019-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anat Benshlomo, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yamamoto M, Ben-Shlomo A, Kameda H, Fukuoka H, Deng N, Ding Y, Melmed S. Somatostatin receptor subtype 5 modifies hypothalamic-pituitary-adrenal axis stress function. JCI Insight. 2018 Oct 4;3(19):e122932. doi: 10.1172/jci.insight.122932. PMID 30282821
- [Background] Altuvia Y, Landgraf P, Lithwick G, Elefant N, Pfeffer S, Aravin A, Brownstein MJ, Tuschl T, Margalit H. Clustering and conservation patterns of human microRNAs. Nucleic Acids Res. 2005 May 12;33(8):2697-706. doi: 10.1093/nar/gki567. Print 2005. PMID 15891114

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexamthesone
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Dexamethesone: Single arm study in which all healthy controls will receive 1 mg of dexamethasone intravenous (IV) injection.
  Dexamethasone 4mg: 1 mg IV dexamethasone will be pushed and miRNA levels will be checked at baseline just before injection and then at 60 minutes after injection.
Arm/Group | Dexamethesone
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 31 [19 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Time of Injection) miRNA Levels and 60 Minutes After Injection
Description: The change of miRNA levels in blood between time of injection (baseline) and 60 minutes after injection. Expressed as miRx ratio: miR expression level normalized to miR7-2-1 expression level and divided by miRx expression at baseline (T0).
Time Frame: Baseline and 60 minutes
Measure: Mean (Standard Deviation); unit: percentage of change
Groups:
- Dexamethesone: Single arm study in which all healthy controls will receive 1 mg of dexamethasone intravenous (IV) injection.
  Dexamethasone 4mg: 1 mg IV dexamethasone will be pushed and miRNA levels will be checked at baseline just before injection and then at 15, 30, 45, and 60 minutes after injection.
Arm/Group | Dexamethesone
Number analyzed (Participants) | 7
percentage of change | 0.939288216 (0.762951729)
Statistical Analysis 1: Comparison: Dexamethesone; Test type: Superiority; p = 0.9, t-test, 2 sided; 2 tailed, unpaired t test with Bonferroni correction; Mean Difference (Final Values) = 0.93928821

ADVERSE EVENTS:
Time Frame: 2.5 months
Arm/Group | Dexamethesone
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/47/NCT04066647/Prot_000.pdf
  • Informed Consent Form (2019-06-25): https://cdn.clinicaltrials.gov/large-docs/47/NCT04066647/ICF_001.pdf